CLINICAL TRIAL: NCT05799937
Title: To Evaluate the Effect of Smoking on Periapical Healing After Non Surgical Root Canal Treatment- a Prospective Cohort Study
Brief Title: Effect of Smoking on Periapical Healing After NSRCT
Status: Completed | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Principal Investigator, Sanjay Tewari, Principal, Postgraduate Institute of Dental Sciences Rohtak
Other Study IDs: PGIDS/BHRC/21/35
Record Dates: First submitted 2021-12-11; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Apical Periodontitis
Keywords: apical periodontitis, periapical pathology, smokers, non-smokers
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group-A Smokers: smoker patients will be recruited in this group
  Interventions: Procedure: Non Surgical Root Canal Treatment
- Group-B Non-Smokers: non smokers or patients who had quit smoking will be recruited in this group
  Interventions: Procedure: Non Surgical Root Canal Treatment

INTERVENTIONS:
Procedure: Non Surgical Root Canal Treatment — After administration of LA and rubber dam isolation, access cavity will be prepared using carbide burs in high speed hand piece with copious irrigation. Working length will be determined using root ZX apex locator and will be verified radiographically. Canal preparation will be done with rotary instruments . 5ml of 5.25% NaOCl will be used as irrigant after each instrument. After instrumentation , the canals will be irrigated with 5.0 ml of 17% EDTA for 1minute followed by irrigation with 5.0 ml of 5.25% NaOCl. Canals will be dried with absorbent paper points, filled with calcium hydroxide paste and access cavity will be restored with IRM. Patients will be recalled after 1 week.At the next appointment, after paste removal, copious irrigation with 5.25% NaOCl will be done and canals will be dried with paper points. Canals will be obturated with Gutta-Percha and ZOE based sealer.

SUMMARY:
Goal of this prospective observational study is determine effect of smoking on periapical healing after NSRCT. Population includes systemically healthy smokers with radiographic evidence of apical periodontitis will be recruited and compared with same type of population of non smokers after non surgical root canal treatment intervention in both the groups. Outcome will be assessed using periapical index scoring system at 6 and 12 months follow up period

DETAILED DESCRIPTION:
The clinical and radiological success of primary non-surgical endodontic treatment in smoker & nonsmoker patients will be compared between both groups and smoking cessation effect on periapical healing will be assessed.

The correlation between the self-reported smoking status & smoking status by urine analysis

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy patients of age 18 years and above, known current smoker patient , a non-smoker or former smoker patient ,should have at least minimum 8 teeth in oral cavity, requiring periapical radiographs of teeth with periapical pathosis

Exclusion Criteria:

* Pregnant or patient having systemic disorders, those patients who are non-compliant and not maintaining oral hygiene, teeth requiring retreatment and having procedural errors. Teeth that are not suitable for rubber dam isolation, teeth that have advanced periodontal disease and having endo-perio lesions and, patients requiring endocarditis prophylaxis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Smokers of age 18 years (male/female) and above having apical periodontitis with age and gender matched controls will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Radiographic healing | 12 months
  Radiographic healing measured by change in ize of apical radiolucency assessed by Periodical index (PAI) .
  PAI score 1 and 2 are classified as healed and PAI score 3,4,and 5 as unhealed.
Clinical Success | 12 month
  Absence of clinical signs and symptoms such as spontaneous pain, presence of sinus tract, swelling, mobility, or sensitivity to percussion or palpation

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sanjay Tewari, MDS, Study Director — Post Graduate Institute Of Dental Sciences,Rohtak
Locations (1):
- PGIDS, Rohtak, Haryana, India